CLINICAL TRIAL: NCT01536002
Title: Pharmacokinetics (PK) of Propofol in Bariatric (Morbidly Obese) Patients
Brief Title: Pharmacokinetics of Propofol in Morbidly Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Tom Heier, Professor, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1.2007.366
Record Dates: First submitted 2012-02-10; First posted 2012-02-20 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Obesity, Morbid
Keywords: Bariatric surgery; Anesthetics, intravenous; Propofol; Pharmacokinetics
MeSH Terms: conditions — Obesity, Morbid | interventions — Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pharmacokinetics (Experimental): Propofol pharmacokinetics
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Intravenous infusion over 30 min of Propofol 3-4 mg/kg body weight
  Other Names: Diprivan

SUMMARY:
The objectives of this study are

* To determine PK of propofol in bariatric patients
* To identify the physiological variables that induce propofol PK changes in bariatric patients, when compared to a normal-weight population.
* To define context-sensitive half-time profiles for propofol in bariatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients admitted to the Aker University Hospital, scheduled for general or bariatric surgery,
* Both genders. Female subjects of childbearing potential must be using adequate contraception (i.e. using oral or IM contraception or an IUCD) and must have a negative pregnancy test (urine beta-HCG).
* Aged 18 - 60 years, both inclusive
* Body mass index (BMI) ≥ 20 kg/m2
* Written informed consent

Exclusion Criteria:

* Patients that are considered not to tolerate a standard dose of propofol administered as a bolus.
* Known hypersensitivity to propofol or its ingredients (soy, lecithin, glycerol, oil acid)
* Known hypersensitivity to any of the anesthetic agents to be used
* Pregnant women
* Lactating women

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2011-06-07 (Actual); Primary Completion 2014-05-07 (Actual); Study Completion 2014-05-07 (Actual)

PRIMARY OUTCOMES:
Propofol plasma concentrations | 0-24 hours
  Arterial blood samples will be collected 0, 1, 2, 4, 8, 10, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 180, 210, 240, 300, 360, 480, 600, 720, and 1440 min after start of propofol bolus infusion. 2 samples will be collected at 0 and 1440 minutes, respectively. The remaining 6 blood samples will be collected according to a block sampling regimen, selected randomly within a time block containing 4 consecutive time points from the time point list noted above. In total 8 samples are drawn from each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Heier, MD,PhD, Principal Investigator — Oslo University Hospital, Oslo, Norway
Locations (1):
- Oslo University Hospital, Oslo, Norway